CLINICAL TRIAL: NCT02099136
Title: Clinical Protocol for a Double-Blind, Placebo-Controlled, Randomized Dose-Ranging Study of Celecoxib (SC-58635) on the Acute Effect of Human UV-Irradiation
Brief Title: Celecoxib in Preventing the Damaging Effects of Sunburn in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2014-00525; NCI-2014-00525 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NQ4-99-02-008 (Other: University of Rochester); N01-CN-85183-Step1 (Other: DCP); N01CN85183 (Other: US NIH Grant/Contract Award Number)
Record Dates: First submitted 2014-03-25; First posted 2014-03-28 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: No Evidence of Disease
MeSH Terms: interventions — Ultraviolet Therapy; Celecoxib; Biopsy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Group I (placebo) (Experimental): Patients receive placebo PO BID for 14 days.
  Interventions: Procedure: UV Light Therapy; Other: Placebo; Procedure: Biopsy; Other: Imaging Biomarker Analysis
- Group II (low-dose celecoxib) (Experimental): Patients receive low-dose celecoxib PO BID for 14 days.
  Interventions: Procedure: UV Light Therapy; Drug: Celecoxib; Procedure: Biopsy; Other: Imaging Biomarker Analysis
- Group III (higher dose celecoxib BID) (Experimental): Patients receive higher dose celecoxib PO BID for 14 days.
  Interventions: Procedure: UV Light Therapy; Drug: Celecoxib; Procedure: Biopsy; Other: Imaging Biomarker Analysis
- Group IV (higher dose celecoxib QD) (Experimental): Patients receive same dose of celecoxib PO as Group III QD for 14 days.
  Interventions: Procedure: UV Light Therapy; Drug: Celecoxib; Procedure: Biopsy; Other: Imaging Biomarker Analysis
- Group V (high-dose celecoxib) (Experimental): Patients receive high-dose celecoxib PO QD for 14 days.
  Interventions: Procedure: UV Light Therapy; Drug: Celecoxib; Procedure: Biopsy; Other: Imaging Biomarker Analysis

INTERVENTIONS:
Procedure: UV Light Therapy — Undergo UV-irradiation
  Other Names: Light Therapy, UV; Therapy, UV Light; Ultraviolet Radiation Therapy
Other: Placebo — Given PO
  Other Names: PLCB
  Arms: Group I (placebo)
Drug: Celecoxib — Given PO
  Other Names: SC-58635
  Arms: Group II (low-dose celecoxib); Group III (higher dose celecoxib BID); Group IV (higher dose celecoxib QD); Group V (high-dose celecoxib)
Procedure: Biopsy — Undergo skin biopsy
  Other Names: Bx
Other: Imaging Biomarker Analysis — Correlative studies

SUMMARY:
This randomized clinical trial studies if celecoxib will prevent the damaging effects of sunburn in healthy volunteers. Exposure to ultraviolet light can induce erythema, sunburn or skin redness caused by inflammation. Celecoxib may reduce skin damage by blocking enzymes associated with sunburn in healthy volunteers. Studying samples of skin in the laboratory from patients receiving ultraviolet-radiation before and after celecoxib treatment may help doctors learn more about the effects celecoxib has on cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Quantify changes in the erythema response in human subjects exposed to minimally erythemic doses of solar-simulated ultraviolet light before and after celecoxib treatment.

II. Determine the effect of celecoxib on various biomarkers following ultraviolet (UV)-irradiation. The modulation of the following biomarkers, before and after treatment with celecoxib are being examined: apoptosis and proliferation indices, prostaglandin E2 (PGE2), cyclooxygenase-1 (COX-1), and cyclooxygenase- 2 (COX-2) levels.

OUTLINE:

Patients undergo UV-irradiation to the right buttock at baseline. Chromameter readings are obtained at 24 hours post UV-irradiation and patients undergo skin biopsy at 24 and 96 hours following UV-irradiation.

Patients are then randomized to 1 of 5 treatment groups.

GROUP I: Patients receive placebo orally (PO) twice daily (BID) for 14 days.

GROUP II: Patients receive low-dose celecoxib PO BID for 14 days.

GROUP III: Patients receive higher dose celecoxib PO BID for 14 days.

GROUP IV: Patients receive same dose of celecoxib PO as Group III once daily (QD) for 14 days.

GROUP V: Patients receive high-dose celecoxib PO QD for 14 days.

After 10 days post-treatment, patients undergo UV-irradiation to the left buttock. Chromameter readings are obtained at 24 hours post UV-irradiation and patients undergo skin biopsy at 24 and 96 hours following UV-irradiation.

After completion of study treatment, patients are followed up at day 25.

ELIGIBILITY:
Inclusion Criteria:

* The subject as Fitzpatrick skin type I, II, or III
* If the subject is female and of childbearing potential (women are considered not of childbearing potential if they are at least 2 years post-menopausal and/or surgically sterile):

  * Has been using adequate contraception (e.g., condom, intrauterine device [IUD], diaphragm and spermicide gel combination) since her last menses and will use adequate contraception during the study, AND
  * Is not lactating, AND
  * Has had a negative pregnancy test (serum or urine) within 14 days prior to the first dose of study medication
* The subject is willing to abstain from the use of non-steroidal anti-inflammatory drugs (NSAIDs) for the duration of the study
* The subject is willing to abstain from the use of all topical agents applied to the buttocks for the duration of the study
* The subject is willing to participate for the duration of the study
* The subject has provided written informed consent prior to administration of any study related procedures

Exclusion Criteria:

* The subject is currently taking any medication that may alter the sunlight response or cause an adverse reaction
* The subject has a history of melanoma, lupus, psoriasis, rosacea, porphyria, photosensitivity disorder, keloid formation, connective tissue disorder, or any disease that would increase the risk associated with study participation
* The subject has excessive hair, blemishes, nevi, uneven pigmentation, sunburn or suntan on the buttocks
* The subject has sun bathed or used a tanning bed to expose the buttocks within 12 months of admission to the study
* The subject has inflammatory bowel disease (e.g., Crohn's disease or ulcerative colitis), a chronic or acute renal or hepatic disorder or a significant coagulation defect or any other condition which in the investigator's opinion might preclude use of an NSAID (e.g., congestive heart failure)
* The subject has an active malignancy of any type or history; subjects who have a history of nonmelanoma skin cancer and have been treated are acceptable; subjects with a history of other malignancies that have been surgically removed and who have no evidence of recurrence for at least five years prior to study enrollment are also acceptable
* The subject has active or suspected peptic ulceration or gastrointestinal bleeding
* The subject has abnormal baseline laboratory test > 1.5 x upper limit of normal (ULN) for serum glutamic oxaloacetic transaminase (SGOT), serum glutamate pyruvate transaminase (SGPT), creatinine, and/or blood urea nitrogen (BUN); all other laboratory abnormalities at baseline thought by the investigator to be clinically significant are also basis for exclusion
* The subject has received any investigational medication within 30 days prior to the first dose of study medication or is scheduled to receive an investigational drug other than celecoxib during the course of this study
* The subject has known hypersensitivity to cyclooxygenase-2 inhibitors, sulfonamides, or NSAIDs
* The subject has been previously admitted to this study
* The subject has significant medical or psychosocial problems that would make the subject a poor candidate, in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 1999-09; Primary Completion 2001-09 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Percent change in erythema | Baseline up to day 25
  Descriptive statistics such as mean, median and standard deviation will be calculated. An increase of 50% in the UV dose needed to reach the minimal erythema dose (MED) will be considered preliminary evidence of drug activity. The modulation of the biomarkers will be compared to the shift in the erythema response. Summary statistics will be provided for plasma drug levels.
Percent change in PGE2 | Baseline up to day 25
  Descriptive statistics such as mean, median and standard deviation will be calculated. An increase of 50% in the UV dose needed to reach the MED will be considered preliminary evidence of drug activity. The modulation of the biomarkers will be compared to the shift in the erythema response. Summary statistics will be provided for plasma drug levels.
Percent change in COX-1 | Baseline up to day 25
  Descriptive statistics such as mean, median and standard deviation will be calculated. An increase of 50% in the UV dose needed to reach the MED will be considered preliminary evidence of drug activity. The modulation of the biomarkers will be compared to the shift in the erythema response. Summary statistics will be provided for plasma drug levels.
Percent change in COX-2 | Baseline up to day 25
  Descriptive statistics such as mean, median and standard deviation will be calculated. An increase of 50% in the UV dose needed to reach the MED will be considered preliminary evidence of drug activity. The modulation of the biomarkers will be compared to the shift in the erythema response. Summary statistics will be provided for plasma drug levels.
Percent change in proliferative index | Baseline up to day 25
  Descriptive statistics such as mean, median and standard deviation will be calculated. An increase of 50% in the UV dose needed to reach the MED will be considered preliminary evidence of drug activity. The modulation of the biomarkers will be compared to the shift in the erythema response. Summary statistics will be provided for plasma drug levels.
Percent change in apoptotic index | Baseline up to day 25
  Descriptive statistics such as mean, median and standard deviation will be calculated. An increase of 50% in the UV dose needed to reach the MED will be considered preliminary evidence of drug activity. The modulation of the biomarkers will be compared to the shift in the erythema response. Summary statistics will be provided for plasma drug levels.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Pentland, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States